CLINICAL TRIAL: NCT01601574
Title: Effects on Glycemic Control and Weight of a Modified Commercial Weight Control Program for People With Type 2 Diabetes
Brief Title: Weight Loss Study for People With Type 2 Diabetes
Acronym: T2D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WW-MUSC-1201
Record Dates: First submitted 2012-04-27; First posted 2012-05-18 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes; Overweight; Obesity
Keywords: Type 2 diabetes; HbA1c; Overweight; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Weight Watchers program (Experimental)
  Interventions: Behavioral: Weight Watchers modified program
- Standard Diabetes Counseling group (Active Comparator)
  Interventions: Other: Standard Care group

INTERVENTIONS:
Behavioral: Weight Watchers modified program — Weight Watchers: For people with Type 2 diabetes including (1) weekly standard in-person Weight Watchers meetings, (2) use of the standard Weight Watchers online program and tools, and (3) two scheduled telephone consultations with a Certified Diabetes Educator (CDE) who will assist the participant in tailoring the standard Weight Watchers program to accommodate the participant's diabetes-related status, with additional unlimited phone and email access to CDEs at the participant's request
  Arms: Modified Weight Watchers program
Other: Standard Care group — One session of in-person diabetic nutritional counseling with a registered dietitian, with follow-up written educational materials.
  Arms: Standard Diabetes Counseling group

SUMMARY:
The purpose of this study is to determine whether the Weight Watchers program modified for use by people with Type 2 diabetes results in more improvements in blood glucose control relative to a control group receiving standard diabetes counseling.

ELIGIBILITY:
Inclusion Criteria:

1. Participant reported diagnosis of Type II diabetes
2. HbA1c between 7%-11% (inclusive)
3. Fasting blood glucose < 240. If a potential participant has a FBG above the inclusion criteria it is acceptable to re-test this potential participant within one week of the original test.
4. BMI 27-50 kg/m2 (inclusive)
5. Age range - 18 - 70 (inclusive)
6. Clearance on medical exam by study physician including EKG
7. No weight loss over the previous 3 months (5kg loss is acceptable with physician discretion)
8. On stable regimen of all medications (including diabetes) for at least 3 months (brief regimens of medications such as antibiotics, steroids, etc. are permitted)
9. All diabetes medications are permitted including insulin.
10. Willing and able to commit to regular physical activity (e.g. walking) five days per week
11. Willingness and ability to make all scheduled appointments required by study protocol
12. Willingness to attend weekly Weight Watchers meetings in the community and to participate in Weight Watchers online program, if so randomized
13. Willing to follow requirements of study protocol
14. Willing and able to provide a valid email address for use in the study
15. Must be able to communicate (oral and written) in English
16. Under the care of a physician for diabetes and willing to give release to contact the MD and request MD's agreement for participant to participate -

Exclusion Criteria:

1. Type 1 Diabetes
2. Cardiovascular/Coronary Heart Disease [e.g., MI or CVA within last 6 months, TIA, clinically significant arrhythmias, uncontrolled hypertension (defined as blood pressure over 160/110); physician's discretion may be more conservative]
3. Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode
4. Taking prescription or OTC weight loss medications within last 4 weeks
5. Currently taking other medications that affect weight (e.g., paroxetine, tricyclics, anti-psychotics)
6. Within the last 4 weeks, use of chromium supplements or any nutrition supplements or herbal products claimed to have a weight loss effect. Participants using other non-excluded nutrition supplements or herbal products must agree to continue at their current level of use throughout the study.
7. Participation in a weight control program within the past 3 months
8. QTc interval >450 msec for males and QTc interval >470 msec for females
9. PHQ-9 total score > 15
10. Thyroid disease for which the participant is untreated or has had treatment changed within the last 6 months. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 6 months is acceptable
11. History of a surgical procedure for weight loss at any time (e.g. gastroplasty, gastric by-pass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve)
12. History of major surgery within three months of enrollment
13. Presence of implanted cardiac defibrillator
14. Orthopedic limitations that would interfere with ability to engage in regular physical activity
15. Gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease
16. Current cancer or cancer treatment, or a history of cancer or cancer treatment within the last 3 years. Persons with successfully resected basal cell carcinoma of the skin may be enrolled if treatment was completed more than 6 months prior to enrollment.
17. History, within the past five years, of clinically diagnosed eating disorders Confidential March 30, 2012 9 including anorexia nervosa or bulimia nervosa.
18. Women who are pregnant, lactating , trying to become pregnant or unwilling to use an effective means of birth control
19. Participation in another clinical trial within 30 days prior to enrollment.
20. Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and unwilling to limit intake to less than 3 drinks per drinking day during study participation
21. Current or past drug abuse
22. Participation in trial by another member of household
23. Hypoglycemic Events:

    a. Evidence of more than 1 severe hypoglycemic event in the past 12 months, unless the participant's treating physician provides written clearance for participation.
24. Any other condition or factor which in the opinion of the study physician or investigator makes it inadvisable for the candidate to participate in the trial -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline and 12 months

SECONDARY OUTCOMES:
Secondary Endpoints | Baseline and 12 months
  Change in weight
Secondary Endpoints | Baseline and 12 months
  Change in BMI
Secondary Endpoints | Baseline and 12 months
  Change in waist circumference
Secondary Endpoints | Baseline and 12 months
  Change in fasting blood glucose
Secondary Endpoints | Baseline and 12 months
  Change in HOMA
Secondary Endpoints | Baseline and 12 months
  Change in cardiovascular risk markers (lipid measures, blood pressure, C-Reactive Protein)
Secondary Endpoints | Baseline and 12 months
  Change in diabetes medications.
Secondary Endpoints | Baseline and 12 months
  Change in various mental health assessments

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M. O'Neil, PhD, Study Director — Medical University of South Carolina
Locations (15):
- United States (15):
  - Diabetes Research and Training Center, University of Alabama at Birmingham, Birmingham, Alabama
  - Scripps Clinical Research, La Jolla, California
  - CSRA Partners in Health, Augusta, Georgia
  - Northwestern University Feinberg School, Chicago, Illinois
  - Obesity Research Center St. Luke's Roosevelt Hospital Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Center for Nutrition and Preventive Medicine, Charlotte, North Carolina
  - Obesity Clinical Trials Program Duke University Medical Center, Durham, North Carolina
  - Your Diabetes Endocrine Nutrition Group Inc., Mentor, Ohio
  - Oregon Weight Loss Surgery, LLC, Portland, Oregon
  - The University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Endocrine Center, Dallas, Texas
  - Oakwell Clinical Research, San Antonio, Texas
  - Washington Center for Weight Management & Research, Inc The Navy League Building, Arlington, Virginia

REFERENCES:
- [Derived] O'Neil PM, Miller-Kovach K, Tuerk PW, Becker LE, Wadden TA, Fujioka K, Hollander PL, Kushner RF, Timothy Garvey W, Rubino DM, Malcolm RJ, Weiss D, Raum WJ, Salyer JL, Hermayer KL, Rost SL, Veliko JL, Sora ND. Randomized controlled trial of a nationally available weight control program tailored for adults with type 2 diabetes. Obesity (Silver Spring). 2016 Nov;24(11):2269-2277. doi: 10.1002/oby.21616. PMID 27804264
- See also: The University of Pennsylvania Center for Weight and Eating Disorders — http://www.med.upenn.edu/weight
- See also: Medical University of South Carolina — http://MUSChealth.com/weight
- See also: Obesity Clinical Trials Program Duke University Medical Center — http://www.dukehealth.org/clinicaltrials
- See also: Comprehensive Weight Control Program Weill Medical College of Cornell University — http://www.weightresearch.net
- See also: Oregon Weight Loss Surgery, LLC — http://www.oregonweightlosssurgery.com
- See also: Scripps Nutrition and Metabolic & Research — http://www.scripps.org/services__clinical-research__active-studies
- See also: University of Alabama at Birmingham Department of Nutrition — http://www.uab.edu/nutrition/
- See also: The Washington Center for Weight Management & Research — http://www.wtmgmt.com
- See also: Baylor Research — http://www.baylorhealth.com/AdvancingMedicine/pages/default.aspx